CLINICAL TRIAL: NCT04794426
Title: Post-operative Pain and Child Behavior of Hall Technique Versus Silver Diamine Fluoride in the Management of Carious Primary Molars: Randomized Clinical Trial
Brief Title: Post-operative Pain and Child Behavior of Hall Technique Versus SDF in the Management of Carious Primary Molars: RCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Noura Mohamed Alhosaini (Other)
Responsible Party: Sponsor-Investigator, Noura Mohamed Alhosaini, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113
Record Dates: First submitted 2021-02-22; First posted 2021-03-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Caries
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (Active Comparator): The group that have caries in primary molars and treat them with Hall Technique
  Interventions: Device: Hall Technique
- experimental group (Experimental): The group that have caries in primary molars and treat them with Silver diamine fluoride (SDF) solution would exert a preventive result in managing early childhood caries ECC.
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Silver diamine fluoride — Previous studies have recommended that Silver diamine fluoride (SDF) solution would exert a preventive result in managing early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention. the objective is useful in arresting early childhood caries (ECC)
  Arms: experimental group
Device: Hall Technique — The first report on the Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique, placed them using a simplified method.
  Arms: control group

SUMMARY:
PICO question:

Papulation: children suffering from caries Intervention: Silver Diamine Fluoride Comparison: Hall technique

Outcome:

Primary Outcome: Intraoperative and postoperative pain Measurement device: Face pain scale Revised8 Measurement unit: Score 0-2-4-6-8-10

Secondary Outcome:

1. Child Anxiety Measurement device: Venham Anxiety rating scale 9 Measurement unit: Six-point scales 0-1-2-3-4-5
2. Child Behavior Measurement device: Venham Behavior rating scale 9 Measurement unit: Six-point scales 0-1-2-3-4-5

DETAILED DESCRIPTION:
Dental caries, also known as tooth decay, it can occur in primary teeth in early childhood, is formed through interaction between acid-producing bacteria and carbohydrate. The caries develops in both the crowns and roots of teeth. Progress of caries depended on the lifestyle of the child (as high numbers of cariogenic bacteria, inadequate salivary flow, insufficient fluoride exposure and poor oral hygiene). To avoid this disease should follow the proper oral hygiene and improve lifestyle 1. A lot of methods found to treatment the decayed tooth - like; Hall technique and Silver diamine fluoride.

The first report on the Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique, placed them using a simplified method2.

Previous studies have recommended that Silver diamine fluoride (SDF) solution would exert a preventive result in managing early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention. the objective is useful in arresting early childhood caries (ECC) 3

ELIGIBILITY:
Inclusion Criteria:

1. Age: From 4 to 6 years
2. Clinical diagnosis of tooth with caries in primary molars within enamel or dentin without pulp disease

Exclusion Criteria:

1. Tooth with signs and symptoms of pulp necrosis
2. Tooth with Root caries
3. Tooth with Spontaneous pain

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-29 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | at 2 days
  Face Pain Scale Revised Immediately after the treatment, any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R). Each child was asked to mark the face that reflected her or his experienced pain during the treatment. The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.
post-operative pain | at 1 week
  Face Pain Scale Revised Immediately after the treatment, any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R). Each child was asked to mark the face that reflected her or his experienced pain during the treatment. The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.
post-operative pain | at 2 weeks
  Face Pain Scale Revised Immediately after the treatment, any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R). Each child was asked to mark the face that reflected her or his experienced pain during the treatment. The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.
post-operative pain | at 1 month
  Face Pain Scale Revised Immediately after the treatment, any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R). Each child was asked to mark the face that reflected her or his experienced pain during the treatment. The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.
post-operative pain | at 6 months
  Face Pain Scale Revised Immediately after the treatment, any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R). Each child was asked to mark the face that reflected her or his experienced pain during the treatment. The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.

SECONDARY OUTCOMES:
Child Anxiety | Immediately
  Venham Anxiety rating scale is a reliable system for rating behavior of children in the dental setting. Six-point scales 0-1-2-3-4-5
Child behavior | Immediately
  Venham behavior rating scale is a reliable system for rating behavior of children in the dental setting. Six-point scales 0-1-2-3-4-5
Intra operative pain | Immediately
  Face Pain Scale Revised Immediately after the treatment, any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R). Each child was asked to mark the face that reflected her or his experienced pain during the treatment. The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B Eltaweil, Prof, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ebrahimi M, Shirazi AS, Afshari E. Success and Behavior During Atraumatic Restorative Treatment, the Hall Technique, and the Stainless Steel Crown Technique for Primary Molar Teeth. Pediatr Dent. 2020 May 15;42(3):187-192. PMID 32522320
- See also: Success and Behavior During Atraumatic Restorative Treatment, the Hall Technique, and the Stainless Steel Crown Technique for Primary Molar Teeth — https://pubmed.ncbi.nlm.nih.gov/32522320/